CLINICAL TRIAL: NCT01838850
Title: A Randomized, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Triple Fixed Dose Combination Therapy With Olmesartan Medoxomil 20mg, Amlodipine 5mg and Hydrochlorothiazide 12.5mg in Patients With Hypertension Not Controlled With Dual Fixed Dose Combination Therapy With Olmesartan Medoxomil 20mg and Hydrochlorothiazide 12.5mg
Brief Title: Efficacy and Safety Study of Olmesartan Medoxomil, Amlodipine and Hydrochlorothiazide Combination Therapy in Patients With Hypertension Not Controlled With Olmesartan Medoxomil and Hydrochlorothiazide Combination Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Korea Co., Ltd., a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS8635-SIT-11-01
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2017-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CS8635 20/5/12.5mg and placebo (Experimental): Participants receiving Olmetec® Plus 20/12.5mg (OM/HCTZ 20/12.5 mg) for the 4-week, Run-in Period but who do not meet their blood pressure goals(Non-responders) could start receiving this triple fixed dose combination therapy (CS8635 20/5/12.5mg (OM/AML/HCTZ 20/5/12.5mg) + placebo) in randomized, 8-week, double-blind Period. The non-responders finishing double-blind treatment could continue the 8-week Open-label Period with CS8635 40/5/12.5mg (OM/AML/HCTZ 40/5/12.5 mg).
  Interventions: Drug: CS8635 20/5/12.5mg and placebo
- Olmetec® Plus 20/12.5mg and placebo (Active Comparator): Participants receiving Olmetec® Plus 20/12.5mg (OM/HCTZ 20/12.5 mg) for the 4-week, Run-in Period but who do not meet their blood pressure goals(Non-responders) could start receiving this dual fixed dose combination therapy (Olmetec® Plus 20/12.5mg (OM/HCTZ 20/12.5mg) + Placebo) in randomized, 8-week, double-blind Period. The non-responders finishing double-blind treatment could continue the 8-week Open-label Period with CS8635 20/5/12.5mg (OM/AML/HCTZ 20/5/12.5 mg).
  Interventions: Drug: Olmetec® Plus 20/12.5mg and placebo

INTERVENTIONS:
Drug: CS8635 20/5/12.5mg and placebo — Run-in period: Coated, Oral tablet containing Olmesartan medoxomil(OM)-Hydrochlorothiazide(HCTZ) 20-12.5mg, given once a day.
  Double-blind period: Coated, Oral tablet containing Olmesartan medoxomil(OM)-Amlodipine (AML)-Hydrochlorothiazide(HCTZ) 20-5-12.5mg, oral placebo tablet. All tablets are given once a day.
  Open-label period: Coated, Oral tablet containing Olmesartan medoxomil(OM)-Amlodipine(AML)-Hydrochlorothiazide(HCTZ) 40-5-12.5mg, given once a day.
  Arms: CS8635 20/5/12.5mg and placebo
Drug: Olmetec® Plus 20/12.5mg and placebo — Run-in period: Coated, Oral tablet containing Olmesartan medoxomil(OM)-Hydrochlorothiazide(HCTZ) 20-12.5mg, given once a day.
  Double-blind period: Coated, Oral tablet containing Olmesartan medoxomil(OM)-Hydrochlorothiazide(HCTZ) 20-12.5mg, oral placebo tablet. All tablets are given once a day.
  Open-label period: Coated, Oral tablet containing Olmesartan medoxomil(OM)-Amlodipine(AML)-Hydrochlorothiazide(HCTZ) 20-5-12.5mg, given once a day.
  Arms: Olmetec® Plus 20/12.5mg and placebo

SUMMARY:
CS-8635 combines three widely prescribed antihypertensive medications, olmesartan medoxomil(OM), amlodipine (AML), and hydrochlorothiazide (HCTZ), to lower blood pressure. The purpose of the study is to evaluate the efficacy and safety of triple therapy with CS-8635 compared with dual therapy in Korean patients with hypertension not controlled with dual fixed dose combination therapy (Olmetec® Plus). The treatments that will be used in this study are as follows: Run-in period -OM/HCTZ 20/12.5 mg (Olmetec® Plus 20/12.5 mg) ; Double blind treatment period - OM/AML/HCTZ 20/5/12.5mg (CS8635 20/5/12.5mg) + its matching placebo vs.OM/HCTZ 20/12.5mg (Olmetec® Plus 20/12.5 mg) + its matching placebo; Open label extension period - OM/AML/HCTZ 40/5/12.5mg (CS8635 40/5/12.5mg) or OM/AML/HCTZ 20/5/12.5mg (CS8635 20/5/12.5mg).

DETAILED DESCRIPTION:
Please refer to arms, outcome measures and eligibility criteria for details.

ELIGIBILITY:
Inclusion Criteria for Screening

* Male or female at the age of 20 to 75 years
* Voluntary written informed consent to participation in this study
* Patients with hypertension either newly diagnosed or without treatment of antihypertensive drugs within 4 weeks of screening, who have mean seated diastolic blood pressure (msDBP) ≥ 100 mmHg at screening, or
* Patients who have been on a stable dose of antihypertensive drugs for at least 4 weeks before run-in period and meet the following blood pressure criteria at screening: Monotherapy: msDBP ≥ 95 mmHg, or Dual combination therapy: msDBP ≥ 90 mmHg, or Triple combination therapy: 70 mmHg ≤ msDBP < 90 mmHg

Inclusion criteria for randomization

* msSBP/DBP at randomization: msSBP ≥ 140 mmHg (msSBP ≥ 130 mmHg in subjects with diabetes or chronic renal disease), and msDBP ≥ 90 mmHg (msDBP ≥ 80 mmHg in subjects with diabetes or chronic renal disease)

Exclusion Criteria:

* msDBP ≥ 115mmHg or msSBP ≥ 200 mmHg measured at screening and randomization
* Patients with mini-max blood pressure difference of SeSBP ≥ 20 mmHg or SeDBP ≥ 10 mmHg in the chosen arm at screening
* Patients with blood pressure difference of SeSBP ≥ 20 mmHg and SeDBP ≥ 10 mmHg in both arms at screening
* Patients with hypersensitivity to the investigational product or any of its components
* Patients with medical history or hypersensitivity to sulfonamide, dihydropyridine, or thiazide diuretics
* History of secondary hypertension or history of any of the diseases suspected of secondary hypertension
* Symptomatic orthostatic hypotension
* Uncontrolled diabetes mellitus
* Severe heart disease, or ischemic heart disease, peripheral vascular disease
* Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter, or other arrhythmia considered clinically significant
* Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, or hemodynamically significant stenosis on aortic valve or mitral valve.
* Severe cerebrovascular disorder
* Known moderate or malignant retinopathy
* Consumption disease , autoimmune disease, or connective tissue disease
* Patients requiring chronic anti-inflammatory treatment
* Anuria or severe renal failure
* Severe hepatic failure, AST or ALT > 3 times the upper limit of normal, biliary obstruction, biliary cirrhosis, or cholestasis
* Patients who have been treated for hyponatremia, hypokalemia, hyperkalemia, hypercalcemia, or symptomatic hyperuricemia
* Addison's disease
* Glucose-galactose malabsorption, galactose intolerance, or Lapp lactase deficiency
* Gastrointestinal tract disease or surgical operation that may affect absorption, distribution, metabolism, and excretion of drugs, presence of active gastritis or gastrointestinal/rectal bleeding considered clinical significant by the investigator, active inflammatory bowel syndrome within the last 12 months, etc
* Patients with history of or suspected of drug or alcohol abuse
* Pregnant or lactating women, or women of childbearing potential who do not agree to use appropriate contraceptive methods such as progestin hormone therapy (Oral, implant), intrauterine device, barrier methods of contraception (condom or occlusive cap (diaphragm or cervical/vault caps) with spermicide), male sterilisation or true abstinence
* Patients who participated in other clinical study within 1 month prior to screening
* Patients considered to be incapable of complying with the protocol

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The changes of seated diastolic blood pressure of the Triple Combinations OM/AML/HCTZ 20/5/12.5mg vs.OM/HCTZ 20/12.5mg | from baseline to week 8

SECONDARY OUTCOMES:
The changes of mean seated systolic blood pressure of the Triple Combinations OM/AML/HCTZ 20/5/12.5mg vs.OM/HCTZ 20/12.5mg | from baseline to Week 8
The changes of mean seated systolic and diastolic blood pressure of the Triple Combinations OM/AML/HCTZ 20/5/12.5mg vs.OM/HCTZ 20/12.5mg | from baseline to week 4
Percentage of subjects achieving blood pressure goal of the Triple Combinations OM/AML/HCTZ 20/5/12.5mg vs.OM/HCTZ 20/12.5mg | at Week 4, and Week 8
Percentage of subjects achieving blood pressure goal of the Triple Combinations OM/AML/HCTZ 40/5/12.5mg vs.OM/AML/HCTZ 20/5/12.5mg | At week 16
The changes of mean seated systolic and diastolic blood pressure of the Triple Combinations OM/AML/HCTZ 40/5/12.5mg vs.OM/AML/HCTZ 20/5/12.5mg | from Week 8 to Week 16

OTHER OUTCOMES:
Collection of safety data from Adverse event, Laboratory test, Physical examination, Vital signs with pulse and ECG | from screening to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Wook Nam, Principal Investigator — Keimyung University Dongsan Medical Center; Cheol-Ho Kim, Principal Investigator — Seoul National University Bundang Hospital; Sang-Hong Baek, Principal Investigator — Seoul St. Mary's Hospital of the Catholic University of Korea; Woo-Baek Chung, Principal Investigator — Yeouido St. Mary's Hospital of the Catholic University of Korea; Woo-Shik Kim, Principal Investigator — Kyunghee University Medical Center; Tae-Hoon Ahn, Principal Investigator — Gachon University Gil Medical Center; Jang-Hyun Cho, Principal Investigator — St. Carollo Hospital; Byung-Hee Oh, Study Chair — Seoul National Univerisity Hospital; Hweung-Kon Hwang, Principal Investigator — Konkuk University Medical Center; Chang-Gyu Park, Principal Investigator — Korea University Guro Hospital; Eun-Seok Shin, Principal Investigator — Ulsan University Hospital; Dong-Ju Choi, Principal Investigator — Seoul National University Bundang Hospital; Joon-Han Shin, Principal Investigator — Ajou University School of Medicine; Myung-Ho Jeong, Principal Investigator — Chonnam National University Hospital; Jin-Ok Jeong, Principal Investigator — Chungnam National University Hospital; Chong-Jin Kim, Principal Investigator — Kyunghee University Hospital at Gandong; Jang-Ho Bae, Principal Investigator — Konyang University Hospital; Seung-Hwan Lee, Principal Investigator — Wonju Severance Christian Hospital; Se-Joong Rim, Principal Investigator — Gangnam Severance Hospital; Jay-Young Rhew, Principal Investigator — Presbyterian medical center; Doo-Il Kim, Principal Investigator — Inje University; Dae-Kyeong Kim, Principal Investigator — Inje University; Soon-Kil Kim, Principal Investigator — Hanyang University; Hye-Sun Seo, Principal Investigator — Soonchunhyang University Hospital; Duk-Hyun Kang, Principal Investigator — Asan Medical Center; Young-Dae Kim, Principal Investigator — Dong-A University Hospital; Dong-Woon Kim, Principal Investigator — Chungbuk National University Hospital; Taek-Jong Hong, Principal Investigator — Pusan National University Hospital; Jong-Won Ha, Principal Investigator — Severance Hospital; Woo-Jung Park, Principal Investigator — Hallym University Medical Center; Tae Ho Kim, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Kee-Sik Kim, Principal Investigator — Daegu Catholic University Medical Center; Seung-Woo Park, Principal Investigator — Sanmsung Medical Center; Wan-Joo Shim, Principal Investigator — Korea University Anam Hospital; Joo-Young Yang, Principal Investigator — Health Insurance Service Ilsan Hospital; Jae-Woong Choi, Principal Investigator — Eulji General Hospital; Sun-Hwa Lee, Principal Investigator — Chonbuk National University Hospital; Jeong-Cheon Ahn, Principal Investigator — Korea University; Keun Lee, Principal Investigator — Seoul Veterans Hospital; Byung-Soo Kim, Principal Investigator — Daedong Hospital
Locations (39):
- South Korea (39):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Medical Center, Anyang
  - Soonchunhyang University Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Daedong Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Presbyterian Medical Center, Cheonju
  - Chonbuk National University Hospital, Cheonju
  - Keimyung University Dongsan Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Konyang University Hospital, Daejeon
  - Health Insurance Service Ilsan Hospital, Goyang
  - Hanyang University Guri Hospital, Guri-si
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Kyunghee University Hospital at Gandong, Seoul
  - Seoul Veterans Hospital, Seoul
  - Sanmsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul St. Mary's Hospital of the Catholic University of Korea, Seoul
  - Asan Medical Center, Seoul
  - Eulji General Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Yeouido St. Mary's Hospital of the Catholic University of Korea, Seoul
  - Korea University Guro Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - St. Carollo Hospital, Suncheon
  - Ajou University Hospital, Suwon
  - Ulsan University hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Sohn IS, Kim CJ, Oh BH, Hong TJ, Park CG, Kim BS, Chung WB; Investigators. Efficacy and Safety Study of Olmesartan Medoxomil, Amlodipine, and Hydrochlorothiazide Combination Therapy in Patients with Hypertension Not Controlled with Olmesartan Medoxomil and Hydrochlorothiazide Combination Therapy: Results of a Randomized, Double-Blind, Multicenter Trial. Am J Cardiovasc Drugs. 2016 Apr;16(2):129-38. doi: 10.1007/s40256-015-0156-x. PMID 26691333